CLINICAL TRIAL: NCT01909804
Title: A Phase 2, Multicenter, Randomized, Open-Label Study to Investigate the Safety and Efficacy of Sofosbuvir + GS-5816 for 12 Weeks in Treatment-Experienced Subjects With Chronic HCV Infection
Brief Title: Safety and Efficacy of Sofosbuvir Plus Velpatasvir With or Without Ribavirin in Treatment-experienced Subjects With Chronic HCV Infection
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Gilead Sciences (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: GS-US-342-0109
Record Dates: First submitted 2013-07-17; First posted 2013-07-29 (Estimated); Results first posted 2016-09-16 (Estimated); Last update posted 2018-11-15 (Actual); Status verified 2016-07

CONDITIONS: Hepatitis C
Keywords: Hepatitis; Genotype 1; Genotype 3; Treatment experienced
MeSH Terms: conditions — Hepatitis C; Hepatitis | interventions — Sofosbuvir; velpatasvir; Ribavirin

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (12):
- SOF+VEL 25 mg (GT3) without cirrhosis (Experimental): Participants with genotype 3 HCV infection without cirrhosis will receive SOF+VEL 25 mg for 12 weeks.
  Interventions: Drug: SOF
- SOF+VEL 25mg+RBV (GT3) without cirrhosis (Experimental): Participants with genotype 3 HCV infection without cirrhosis will receive SOF+VEL 25 mg plus RBV for 12 weeks.
  Interventions: Drug: SOF; Drug: VEL; Drug: RBV
- SOF+VEL 100 mg (GT3) without cirrhosis (Experimental): Participants with genotype 3 HCV infection without cirrhosis will receive SOF+VEL 100 mg for 12 weeks.
  Interventions: Drug: SOF; Drug: VEL
- SOF+VEL 100 mg+RBV (GT3) without cirrhosis (Experimental): Participants with genotype 3 HCV infection without cirrhosis will receive SOF+VEL 100 mg plus RBV for 12 weeks.
  Interventions: Drug: SOF; Drug: VEL; Drug: RBV
- SOF+VEL 25 mg (GT3) with cirrhosis (Experimental): Participants with genotype 3 HCV infection with cirrhosis will receive SOF+VEL 25 mg for 12 weeks.
  Interventions: Drug: SOF; Drug: VEL
- SOF+VEL 25 mg+RBV (GT3) with cirrhosis (Experimental): Participants with genotype 3 HCV infection with cirrhosis will receive SOF+VEL 25 mg plus RBV for 12 weeks.
  Interventions: Drug: SOF; Drug: RBV
- SOF+VEL 100 mg (GT3) with cirrhosis (Experimental): Participants with genotype 3 HCV infection with cirrhosis will receive SOF+VEL 100 mg for 12 weeks.
  Interventions: Drug: SOF; Drug: VEL
- SOF+VEL 100 mg+RBV (GT3) with cirrhosis (Experimental): Participants with genotype 3 HCV infection with cirrhosis will receive SOF+VEL 100 mg plus RBV for 12 weeks.
  Interventions: Drug: SOF; Drug: VEL; Drug: RBV
- SOF+VEL 25 mg (GT1) (Experimental): Participants with genotype 1 HCV infection will receive SOF+VEL 25 mg for 12 weeks.
  Interventions: Drug: SOF; Drug: VEL
- SOF+VEL 25 mg+RBV (GT1) (Experimental): Participants with genotype 1 HCV infection will receive SOF+VEL 25 mg plus RBV for 12 weeks.
  Interventions: Drug: SOF; Drug: VEL; Drug: RBV
- SOF+VEL 100 mg (GT1) (Experimental): Participants with genotype 1 HCV infection will receive SOF+VEL 100 mg for 12 weeks.
  Interventions: Drug: SOF; Drug: VEL
- SOF+VEL 100 mg+RBV (GT1) (Experimental): Participants with genotype 1 HCV infection will receive SOF+VEL 100 mg plus RBV for 12 weeks.
  Interventions: Drug: SOF; Drug: VEL; Drug: RBV

INTERVENTIONS:
Drug: SOF — 400 mg tablet administered orally once daily
  Other Names: Sovaldi®; GS-7977; PSI-7977
Drug: VEL — Tablet administered orally once daily
  Other Names: GS-5816
  Arms: SOF+VEL 100 mg (GT1); SOF+VEL 100 mg (GT3) with cirrhosis; SOF+VEL 100 mg (GT3) without cirrhosis; SOF+VEL 100 mg+RBV (GT1); SOF+VEL 100 mg+RBV (GT3) with cirrhosis; SOF+VEL 100 mg+RBV (GT3) without cirrhosis; SOF+VEL 25 mg (GT1); SOF+VEL 25 mg (GT3) with cirrhosis; SOF+VEL 25 mg+RBV (GT1); SOF+VEL 25mg+RBV (GT3) without cirrhosis
Drug: RBV — 200 mg tablets administered orally in a divided daily dose according to package insert weight-based dosing recommendations (< 75 kg = 1000 mg and ≥ 75 kg = 1200 mg)
  Other Names: Ribasphere®
  Arms: SOF+VEL 100 mg+RBV (GT1); SOF+VEL 100 mg+RBV (GT3) with cirrhosis; SOF+VEL 100 mg+RBV (GT3) without cirrhosis; SOF+VEL 25 mg+RBV (GT1); SOF+VEL 25 mg+RBV (GT3) with cirrhosis; SOF+VEL 25mg+RBV (GT3) without cirrhosis

SUMMARY:
The primary objectives of this study are to evaluate the antiviral efficacy, safety, and tolerability of sofosbuvir (SOF) + velpatasvir (VEL; GS-5816) with or without ribavirin (RBV) in treatment-naive adults with chronic genotype (GT) 1 or 3 hepatitis C virus (HCV) infection.

ELIGIBILITY:
Inclusion Criteria:

* Body mass index (BMI) ≥ 18 kg/m^2
* HCV RNA ≥ 10000 IU/mL at screening
* Prior treatment failure to a regimen including interferon with or without RBV
* HCV genotype 1 or 3
* Chronic HCV infection
* Cirrhosis determination
* Use of highly effective contraception methods if female of childbearing potential or sexually active male

Exclusion Criteria:

* Current or prior history of clinically significant illness other than HCV
* Screening ECG with clinically significant abnormalities
* Prior exposure to HCV specific direct acting antiviral agent
* Pregnant or nursing female or male with pregnant female partner
* Chronic liver disease of non-HCV etiology
* Hepatitis B
* Active drug abuse
* Use of any prohibited concomitant medications

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 323 (Actual)
Dates: Start 2013-06; Primary Completion 2014-05 (Actual); Study Completion 2014-08 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: John McNally, Study Director — Gilead Sciences
Locations (49):
- United States (40):
  - Long Beach, California
  - Los Angeles, California
  - Pasadena, California
  - San Diego, California
  - Denver, Colorado
  - Gainesville, Florida
  - Jacksonville, Florida
  - Miami, Florida
  - Orlando, Florida
  - Tampa, Florida
  - Wellington, Florida
  - Atlanta, Georgia
  - Marietta, Georgia
  - Chicago, Illinois
  - Indianapolis, Indiana
  - Baltimore, Maryland
  - Boston, Massachusetts
  - Detroit, Michigan
  - Hillsborough, New Jersey
  - Santa Fe, New Mexico
  - Great Neck, New York
  - New York, New York
  - Asheville, North Carolina
  - Durham, North Carolina
  - Fayetteville, North Carolina
  - Winston-Salem, North Carolina
  - Portland, Oregon
  - Philadelphia, Pennsylvania
  - Pittsburgh, Pennsylvania
  - Providence, Rhode Island
  - Germantown, Tennessee
  - Nashville, Tennessee
  - Arlington, Texas
  - Dallas, Texas
  - San Antonio, Texas
  - Annandale, Virginia
  - Fairfax, Virginia
  - Newport News, Virginia
  - Norfolk, Virginia
  - Seattle, Washington
- Australia (6):
  - Camperdown, New South Wales
  - Darlinghurst, New South Wales
  - Clayton, Victoria
  - Melbourne, Victoria
  - Fremantle, Western Australia
  - Perth, Western Australia
- New Zealand (2):
  - Auckland
  - Christchurch
- San Juan, Puerto Rico

IPD SHARING:
Plan to Share IPD: Yes
Qualified external researchers may request IPD for this study after study completion. For more information, please visit our website at http://www.gilead.com/research/disclosure-and-transparency.
Supporting Information: Study Protocol, SAP
Time Frame: 18 months after study completion
Access Criteria: A secured external environment with username, password, and RSA code.
URL: http://www.gilead.com/research/disclosure-and-transparency

REFERENCES:
- [Result] Pianko S, Flamm SL, Shiffman ML, Kumar S, Strasser SI, Dore GJ, et al. High Efficacy of Treatment with Sofosbuvir+GS-5816±Ribavirin for 12 Weeks in Treatment-Experienced Patients with Genotype 1 or 3 HCV Infection [Abstract 197]. American Association for the Study of Liver Diseases (AASLD); 2014 November 7-11; Boston MA United States.
- [Result] Pianko S, Flamm SL, Shiffman ML, Kumar S, Strasser SI, Dore GJ, McNally J, Brainard DM, Han L, Doehle B, Mogalian E, McHutchison JG, Rabinovitz M, Towner WJ, Gane EJ, Stedman CA, Reddy KR, Roberts SK. Sofosbuvir Plus Velpatasvir Combination Therapy for Treatment-Experienced Patients With Genotype 1 or 3 Hepatitis C Virus Infection: A Randomized Trial. Ann Intern Med. 2015 Dec 1;163(11):809-17. doi: 10.7326/M15-1014. Epub 2015 Nov 10. PMID 26551263

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants were enrolled at study sites in Australia, New Zealand, and the United States. The first participant was screened on 17 June 2013. The last study visit occurred on 22 August 2014.
Pre-assignment Details: 416 participants were screened.
Groups:
- SOF+VEL 25 mg (GT3 Non-Cirrhotic): Sofosbuvir (SOF) 400 mg tablet + VEL 25 mg tablet administered orally once daily for 12 weeks (genotype (GT) 3 non-cirrhotic)
- SOF+VEL 25 mg + RBV (GT3 Non-Cirrhotic): SOF 400 mg tablet + velpatasvir (VEL) 25 mg tablet administered orally once daily + ribavirin (RBV) tablets (1000 or 1200 mg daily based on weight) for 12 weeks (genotype 3 non-cirrhotic)
- SOF+VEL 100 mg (GT3 Non-Cirrhotic): SOF 400 mg tablet + VEL 100 mg tablet administered orally once daily for 12 weeks (genotype 3 non-cirrhotic)
- SOF+VEL 100 mg + RBV (GT3 Non-Cirrhotic): SOF 400 mg tablet + VEL 100 mg tablet administered orally once daily + RBV tablets (1000 or 1200 mg daily based on weight) for 12 weeks (genotype 3 non-cirrhotic)
- SOF+VEL 25 mg (GT3 Cirrhotic): SOF 400 mg tablet + VEL 25 mg tablet administered orally once daily for 12 weeks (genotype 3 cirrhotic)
- SOF+VEL 25 mg + RBV (GT3 Cirrhotic): SOF 400 mg tablet + VEL 25 mg tablet administered orally once daily + RBV tablets (1000 or 1200 mg daily based on weight) for 12 weeks (genotype 3 cirrhotic)
- SOF+VEL 100 mg (GT3 Cirrhotic): SOF 400 mg tablet + VEL 100 mg tablet administered orally once daily for 12 weeks (genotype 3 cirrhotic)
- SOF+VEL 100 mg + RBV (GT3 Cirrhotic): SOF 400 mg tablet + VEL 100 mg tablet administered orally once daily + RBV tablets (1000 or 1200 mg daily based on weight) for 12 weeks (genotype 3 cirrhotic)
- SOF+VEL 25 mg (GT1): SOF 400 mg tablet + VEL 25 mg tablet administered orally once daily for 12 weeks (genotype 1)
- SOF+VEL 25 mg + RBV (GT1): SOF 400 mg tablet + VEL 25 mg tablet administered orally once daily + RBV tablets (1000 or 1200 mg daily based on weight) for 12 weeks (genotype 1)
- SOF+VEL 100 mg (GT1): SOF 400 mg tablet + VEL 100 mg tablet administered orally once daily for 12 weeks (genotype 1)
- SOF+VEL 100 mg + RBV (GT1): SOF 400 mg tablet + VEL 100 mg tablet administered orally once daily + RBV tablets (1000 or 1200 mg daily based on weight) for 12 weeks (genotype 1)
Period: Overall Study
Arm/Group | SOF+VEL 25 mg (GT3 Non-Cirrhotic) | SOF+VEL 25 mg + RBV (GT3 Non-Cirrhotic) | SOF+VEL 100 mg (GT3 Non-Cirrhotic) | SOF+VEL 100 mg + RBV (GT3 Non-Cirrhotic) | SOF+VEL 25 mg (GT3 Cirrhotic) | SOF+VEL 25 mg + RBV (GT3 Cirrhotic) | SOF+VEL 100 mg (GT3 Cirrhotic) | SOF+VEL 100 mg + RBV (GT3 Cirrhotic) | SOF+VEL 25 mg (GT1) | SOF+VEL 25 mg + RBV (GT1) | SOF+VEL 100 mg (GT1) | SOF+VEL 100 mg + RBV (GT1)
Started | 26 | 28 | 27 | 26 | 26 | 25 | 27 | 26 | 27 | 29 | 27 | 29
Completed | 22 | 27 | 27 | 26 | 18 | 21 | 25 | 25 | 27 | 28 | 26 | 26
Not Completed | 4 | 1 | 0 | 0 | 8 | 4 | 2 | 1 | 0 | 1 | 1 | 3
Not completed — Randomized but Never Treated | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 1
Not completed — Death | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Not completed — Lack of Efficacy | 4 | 1 | 0 | 0 | 7 | 3 | 1 | 1 | 0 | 1 | 0 | 1
Not completed — Withdrew Consent | 0 | 0 | 0 | 0 | 1 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Not completed — Protocol Violation | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1

BASELINE CHARACTERISTICS:
Population: Safety Analysis Set: participants who were randomized and received at least 1 dose of study drug.
Groups:
- SOF+VEL 25 mg (GT3 Non-Cirrhotic): SOF 400 mg tablet + VEL 25 mg tablet administered orally once daily for 12 weeks (genotype (GT) 3 non-cirrhotic)
- SOF+VEL 25 mg + RBV (GT3 Non-Cirrhotic): SOF 400 mg tablet + VEL 25 mg tablet administered orally once daily + RBV tablets (1000 or 1200 mg daily based on weight) for 12 weeks (genotype 3 non-cirrhotic)
- Total: Total of all reporting groups
Arm/Group | SOF+VEL 25 mg (GT3 Non-Cirrhotic) | SOF+VEL 25 mg + RBV (GT3 Non-Cirrhotic) | SOF+VEL 100 mg (GT3 Non-Cirrhotic) | SOF+VEL 100 mg + RBV (GT3 Non-Cirrhotic) | SOF+VEL 25 mg (GT3 Cirrhotic) | SOF+VEL 25 mg + RBV (GT3 Cirrhotic) | SOF+VEL 100 mg (GT3 Cirrhotic) | SOF+VEL 100 mg + RBV (GT3 Cirrhotic) | SOF+VEL 25 mg (GT1) | SOF+VEL 25 mg + RBV (GT1) | SOF+VEL 100 mg (GT1) | SOF+VEL 100 mg + RBV (GT1) | Total
Number analyzed (Participants) | 26 | 28 | 27 | 26 | 26 | 25 | 26 | 26 | 27 | 29 | 27 | 28 | 321
Age, Continuous [Mean (Standard Deviation); unit: years] | 54 (11.8) | 51 (10.4) | 55 (6.9) | 56 (6.4) | 57 (7.0) | 56 (5.6) | 56 (5.7) | 54 (4.7) | 55 (8.1) | 57 (5.8) | 57 (6.4) | 56 (6.0) | 55 (7.4)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 8 | 6 | 9 | 9 | 5 | 10 | 6 | 6 | 12 | 7 | 12 | 10 | 100
  Male | 18 | 22 | 18 | 17 | 21 | 15 | 20 | 20 | 15 | 22 | 15 | 18 | 221
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 1 | 2 | 1 | 2 | 1 | 1 | 2 | 0 | 2 | 1 | 4 | 3 | 20
  Not Hispanic or Latino | 25 | 26 | 26 | 24 | 25 | 24 | 24 | 26 | 25 | 28 | 23 | 25 | 301
  Unknown or Not Reported | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Race/Ethnicity, Customized [Number; unit: participants]
  American Indian or Alaska Native | 0 | 0 | 1 | 1 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 1 | 4
  Asian | 1 | 1 | 1 | 0 | 1 | 2 | 0 | 1 | 0 | 0 | 0 | 2 | 9
  Black or African American | 0 | 1 | 0 | 1 | 0 | 0 | 0 | 0 | 7 | 2 | 4 | 4 | 19
  Native Hawaiian or Pacific Islander | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 1
  White | 25 | 26 | 25 | 24 | 25 | 23 | 25 | 24 | 20 | 27 | 23 | 21 | 288
HCV Genotype [Number; unit: participants]
  Genotype 1a | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 19 | 22 | 21 | 22 | 84
  Genotype 1b | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 7 | 7 | 6 | 6 | 26
  Genotype 1 (no confirmed subtype) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 1
  Genotype 3 | 26 | 28 | 27 | 26 | 26 | 25 | 26 | 26 | 0 | 0 | 0 | 0 | 210
IL28b Status [Number; unit: participants] — CC, CT, and TT alleles are different forms of the IL28b gene.
  participants
    CC | 8 | 10 | 8 | 11 | 12 | 5 | 12 | 13 | 0 | 1 | 2 | 3 | 85
    CT | 16 | 14 | 13 | 12 | 11 | 14 | 11 | 10 | 19 | 21 | 17 | 19 | 177
    TT | 2 | 4 | 6 | 3 | 3 | 6 | 3 | 3 | 8 | 7 | 8 | 6 | 59
Cirrhosis Status [Number; unit: participants]
  Absent | 25 | 27 | 27 | 24 | 0 | 0 | 0 | 0 | 17 | 19 | 18 | 18 | 175
  Present | 0 | 0 | 0 | 0 | 26 | 25 | 26 | 26 | 8 | 10 | 7 | 10 | 138
  Missing | 1 | 1 | 0 | 2 | 0 | 0 | 0 | 0 | 2 | 0 | 2 | 0 | 8
HCV RNA [Mean (Standard Deviation); unit: log10 IU/mL] | 6.7 (0.76) | 6.6 (0.70) | 6.6 (0.59) | 6.7 (0.53) | 6.6 (0.46) | 6.2 (0.68) | 6.4 (0.76) | 6.7 (0.51) | 6.5 (0.59) | 6.8 (0.37) | 6.4 (0.53) | 6.5 (0.43) | 6.6 (0.60)
HCV RNA Category [Number; unit: participants]
  < 800,000 IU/mL | 5 | 6 | 2 | 2 | 3 | 7 | 7 | 2 | 6 | 0 | 3 | 3 | 46
  ≥ 800,000 IU/mL | 21 | 22 | 25 | 24 | 23 | 18 | 19 | 24 | 21 | 29 | 24 | 25 | 275
Prior HCV Treatment [Number; unit: participants]
  Non-responder | 7 | 10 | 7 | 5 | 6 | 9 | 10 | 3 | 6 | 13 | 7 | 8 | 91
  Relapse / Breakthrough | 19 | 18 | 20 | 21 | 20 | 16 | 16 | 23 | 21 | 16 | 20 | 20 | 230

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Participants With Sustained Virologic Response (SVR) 12 Weeks After Discontinuation of Therapy (SVR12)
Description: SVR12 was defined as HCV RNA < the lower limit of quantitation (LLOQ; ie, 15 IU/mL) at 12 weeks after stopping study treatment.
Time Frame: Posttreatment Week 12
Population: Full Analysis Set: participants randomized into the study and received at least 1 dose of study drug.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | SOF+VEL 25 mg (GT3 Non-Cirrhotic) | SOF+VEL 25 mg + RBV (GT3 Non-Cirrhotic) | SOF+VEL 100 mg (GT3 Non-Cirrhotic) | SOF+VEL 100 mg + RBV (GT3 Non-Cirrhotic) | SOF+VEL 25 mg (GT3 Cirrhotic) | SOF+VEL 25 mg + RBV (GT3 Cirrhotic) | SOF+VEL 100 mg (GT3 Cirrhotic) | SOF+VEL 100 mg + RBV (GT3 Cirrhotic) | SOF+VEL 25 mg (GT1) | SOF+VEL 25 mg + RBV (GT1) | SOF+VEL 100 mg (GT1) | SOF+VEL 100 mg + RBV (GT1)
Number analyzed (Participants) | 26 | 28 | 27 | 26 | 26 | 25 | 26 | 26 | 27 | 29 | 27 | 28
percentage of participants | 84.6 [65.1 to 95.6] | 96.4 [81.7 to 99.9] | 100.0 [87.2 to 100.0] | 100.0 [86.8 to 100.0] | 57.7 [36.9 to 76.6] | 84.0 [63.9 to 95.5] | 88.5 [69.8 to 97.6] | 96.2 [80.4 to 99.9] | 100.0 [87.2 to 100.0] | 96.6 [82.2 to 99.9] | 100.0 [87.2 to 100.0] | 96.4 [81.7 to 99.9]

2. Primary Outcome: Percentage of Participants Who Permanently Discontinued Any Study Drug Due to an Adverse Event
Time Frame: Up to 12 weeks
Population: Safety Analysis Set
Measure: Number; unit: percentage of participants
Groups:
- SOF+VEL 25 mg: SOF 400 mg tablet + VEL 25 mg tablet administered orally once daily for 12 weeks (genotypes 1 and 3)
- SOF+VEL 25 mg + RBV: SOF 400 mg tablet + VEL 25 mg tablet administered orally once daily + RBV tablets (1000 or 1200 mg daily based on weight) for 12 weeks (genotypes 1 and 3)
- SOF+VEL 100 mg: SOF 400 mg tablet + VEL 100 mg tablet administered orally once daily for 12 weeks (genotypes 1 and 3)
- SOF+VEL 100 mg + RBV: SOF 400 mg tablet + VEL 100 mg tablet administered orally once daily + RBV tablets (1000 or 1200 mg daily based on weight) for 12 weeks (genotypes 1 and 3)
Arm/Group | SOF+VEL 25 mg | SOF+VEL 25 mg + RBV | SOF+VEL 100 mg | SOF+VEL 100 mg + RBV
Number analyzed (Participants) | 79 | 82 | 80 | 80
percentage of participants | 0 | 1.2 | 0 | 0

3. Secondary Outcome: Percentage of Participants With SVR at 4 and 24 Weeks After Discontinuation of Therapy (SVR4 and SVR24)
Description: SVR4 and SVR 24 were defined as HCV RNA < LLOQ at 4 and 24 weeks after stopping study treatment, respectively.
Time Frame: Posttreatment Weeks 4 and 24
Population: Full Analysis Set
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | SOF+VEL 25 mg (GT3 Non-Cirrhotic) | SOF+VEL 25 mg + RBV (GT3 Non-Cirrhotic) | SOF+VEL 100 mg (GT3 Non-Cirrhotic) | SOF+VEL 100 mg + RBV (GT3 Non-Cirrhotic) | SOF+VEL 25 mg (GT3 Cirrhotic) | SOF+VEL 25 mg + RBV (GT3 Cirrhotic) | SOF+VEL 100 mg (GT3 Cirrhotic) | SOF+VEL 100 mg + RBV (GT3 Cirrhotic) | SOF+VEL 25 mg (GT1) | SOF+VEL 25 mg + RBV (GT1) | SOF+VEL 100 mg (GT1) | SOF+VEL 100 mg + RBV (GT1)
Number analyzed (Participants) | 26 | 28 | 27 | 26 | 26 | 25 | 26 | 26 | 27 | 29 | 27 | 28
percentage of participants
  SVR4 | 88.5 [69.8 to 97.6] | 96.4 [81.7 to 99.9] | 100.0 [87.2 to 100.0] | 100.0 [86.8 to 100.0] | 61.5 [40.6 to 79.8] | 84.0 [63.9 to 95.5] | 88.5 [69.8 to 97.6] | 96.2 [80.4 to 99.9] | 100.0 [87.2 to 100.0] | 96.6 [82.2 to 99.9] | 100.0 [87.2 to 100.0] | 96.4 [81.7 to 99.9]
  SVR24 | 84.6 [65.1 to 95.6] | 96.4 [81.7 to 99.9] | 100.0 [87.2 to 100.0] | 100.0 [86.8 to 100.0] | 57.7 [36.9 to 76.6] | 84.0 [63.9 to 95.5] | 92.3 [74.9 to 99.1] | 96.2 [80.4 to 99.9] | 100.0 [87.2 to 100.0] | 96.6 [82.2 to 99.9] | 100.0 [87.2 to 100.0] | 96.4 [81.7 to 99.9]

4. Secondary Outcome: Percentage of Participants With Virologic Failure
Description: Virologic failure was defined as:
  * On-treatment virologic failure:
    * Breakthrough (confirmed HCV RNA ≥ LLOQ after having previously had HCV RNA < LLOQ while on treatment), or
    * Rebound (confirmed > 1 log10 IU/mL increase in HCV RNA from nadir while on treatment), or
    * Non-response (HCV RNA persistently ≥ LLOQ through 8 weeks of treatment)
  * Virologic relapse:
    * Confirmed HCV RNA ≥ LLOQ during the posttreatment period having achieved HCV RNA < LLOQ at last on-treatment visit.
Time Frame: Up to Posttreatment Week 24
Population: Full Analysis Set
Measure: Number; unit: percentage of participants
Arm/Group | SOF+VEL 25 mg (GT3 Non-Cirrhotic) | SOF+VEL 25 mg + RBV (GT3 Non-Cirrhotic) | SOF+VEL 100 mg (GT3 Non-Cirrhotic) | SOF+VEL 100 mg + RBV (GT3 Non-Cirrhotic) | SOF+VEL 25 mg (GT3 Cirrhotic) | SOF+VEL 25 mg + RBV (GT3 Cirrhotic) | SOF+VEL 100 mg (GT3 Cirrhotic) | SOF+VEL 100 mg + RBV (GT3 Cirrhotic) | SOF+VEL 25 mg (GT1) | SOF+VEL 25 mg + RBV (GT1) | SOF+VEL 100 mg (GT1) | SOF+VEL 100 mg + RBV (GT1)
Number analyzed (Participants) | 26 | 28 | 27 | 26 | 26 | 25 | 26 | 26 | 27 | 29 | 27 | 28
percentage of participants | 15.4 | 3.6 | 0 | 0 | 42.3 | 12.0 | 11.5 | 3.8 | 0 | 3.4 | 0 | 3.6

ADVERSE EVENTS:
Time Frame: Up to 12 weeks plus 30 days
Description: Safety Analysis Set
Arm/Group | SOF+VEL 25 mg | SOF+VEL 25 mg + RBV | SOF+VEL 100 mg | SOF+VEL 100 mg + RBV
Serious Adverse Events (participants affected / at risk) | 1/79 | 0/82 | 4/80 | 3/80
Other Adverse Events (participants affected / at risk) | 54/79 | 61/82 | 54/80 | 62/80
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | SOF+VEL 25 mg (N=79) | SOF+VEL 25 mg + RBV (N=82) | SOF+VEL 100 mg (N=80) | SOF+VEL 100 mg + RBV (N=80)
Acute myocardial infarction (Cardiac disorders) | 0 | 0 | 0 | 1
Atrial fibrillation (Cardiac disorders) | 0 | 0 | 1 | 0
Abdominal pain (Gastrointestinal disorders) | 0 | 0 | 0 | 1
Drug withdrawal syndrome (General disorders) | 0 | 0 | 0 | 1
Thrombosis in device (General disorders) | 0 | 0 | 1 | 0
Viral infection (Infections and infestations) | 1 | 0 | 0 | 0
Hypersensitivity vasculitis (Skin and subcutaneous tissue disorders) | 0 | 0 | 1 | 0
Hypertension (Vascular disorders) | 0 | 0 | 1 | 0
May-Thurner syndrome (Vascular disorders) | 0 | 0 | 1 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | SOF+VEL 25 mg (N=79) | SOF+VEL 25 mg + RBV (N=82) | SOF+VEL 100 mg (N=80) | SOF+VEL 100 mg + RBV (N=80)
Anaemia (Blood and lymphatic system disorders) | 0 | 4 | 0 | 5
Constipation (Gastrointestinal disorders) | 4 | 3 | 4 | 6
Diarrhoea (Gastrointestinal disorders) | 9 | 4 | 9 | 4
Dyspepsia (Gastrointestinal disorders) | 2 | 3 | 4 | 6
Gastrooesophageal reflux disease (Gastrointestinal disorders) | 4 | 2 | 1 | 4
Nausea (Gastrointestinal disorders) | 12 | 18 | 7 | 18
Vomiting (Gastrointestinal disorders) | 1 | 4 | 1 | 4
Fatigue (General disorders) | 16 | 27 | 19 | 27
Influenza like illness (General disorders) | 0 | 1 | 4 | 1
Nasopharyngitis (Infections and infestations) | 1 | 2 | 2 | 4
Upper respiratory tract infection (Infections and infestations) | 6 | 7 | 5 | 3
Laceration (Injury, poisoning and procedural complications) | 0 | 2 | 1 | 4
Decreased appetite (Metabolism and nutrition disorders) | 4 | 3 | 1 | 2
Arthralgia (Musculoskeletal and connective tissue disorders) | 3 | 4 | 7 | 3
Back pain (Musculoskeletal and connective tissue disorders) | 3 | 6 | 3 | 2
Muscle spasms (Musculoskeletal and connective tissue disorders) | 2 | 1 | 1 | 4
Myalgia (Musculoskeletal and connective tissue disorders) | 1 | 4 | 6 | 4
Dizziness (Nervous system disorders) | 7 | 8 | 1 | 4
Headache (Nervous system disorders) | 23 | 28 | 18 | 24
Insomnia (Psychiatric disorders) | 12 | 11 | 6 | 16
Irritability (Psychiatric disorders) | 6 | 6 | 3 | 12
Cough (Respiratory, thoracic and mediastinal disorders) | 5 | 5 | 4 | 7
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 0 | 6 | 1 | 5
Dyspnoea exertional (Respiratory, thoracic and mediastinal disorders) | 0 | 3 | 0 | 5
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 4 | 1 | 0 | 0
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 4 | 5 | 1 | 1
Dry skin (Skin and subcutaneous tissue disorders) | 1 | 6 | 1 | 1
Pruritus (Skin and subcutaneous tissue disorders) | 2 | 9 | 2 | 12
Rash (Skin and subcutaneous tissue disorders) | 4 | 5 | 2 | 9

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
After conclusion of the study and without prior written approval from Gilead, investigators in this study may communicate, orally present, or publish in scientific journals or other media only after the following conditions have been met:

* The results of the study in their entirety have been publicly disclosed by or with the consent of Gilead in an abstract, manuscript, or presentation form; or
* The study has been completed at all study sites for at least 2 years